CLINICAL TRIAL: NCT03923400
Title: Characteristics and Prognosis of Jejunoileal Gastrointestinal Stromal Tumors (GISTs) in the Era of Imatinib. A Comparative Retrospective Study With Gastric GISTs.
Brief Title: Jejunoileal vs Gastric GIST in the Era of Imatinib.
Status: Completed | Type: Observational
Sponsor: Hospital Universitario Virgen de la Arrixaca (Other)
Responsible Party: Principal Investigator, David Ferreras, Principal Investigator, Hospital Universitario Virgen de la Arrixaca
Other Study IDs: YiGi
Record Dates: First submitted 2019-03-26; First posted 2019-04-22 (Actual); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Disease-free Survival; Overall Survival; Recurrence
Keywords: GIST; small bowel; jejunum; ileum
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- JI-GIST: The series comprises 77 patients, of which 29 (37.7%) were located in the jejunum or ileum (JI-GIST).
- G-GIST: The series comprises 77 patients, of which 48 (62.3%) were located in the stomach (G-GIST).

SUMMARY:
Introduction: Gastrointestinal Stromal Tumors (GISTs) located in the jejunum or ileum (JI-GIST) are considered of worse prognosis compared to other locations. It has been suggested that this dogma should be revised. The aim of this study is to describe the characteristics of jejunoileal GISTs and its prognosis; and to compare them with gastric GISTs in the era of imatinib.

Patients and methods: We retrospectively reviewed the clinical histories of all the patients diagnosed with GISTs between January 2000 and November 2016. Clinical and pathological data, as well recurrence, metastatic, disease-free survival (DFS) as overall (OS) rates of patients with JI-GIST or gastric GIST (G-GIST) were collected and compared.

ELIGIBILITY:
Inclusion Criteria:

* Any kind of primary mesenchymal tumor of the gastrointestinal tract with a histomorphological and immunohistochemical (CD117 (+) and/or DOG1 (+)) profile consistent with GIST.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: GIST diagnosis was established by an experienced board-certified pathologist who reviewed our database prospectively maintained. After revision, we included in the study any kind of primary mesenchymal tumor of the gastrointestinal tract with a histomorphological and immunohistochemical (CD117 (+) and/or DOG1 (+)) profile consistent with GIST. The patients were divided into two groups: patients with GISTs located in the jejunum or ileum, comprising the JI-GIST group; and patients with gastric GISTs, comprising the G-GIST group.
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2017-01-31 (Actual)

PRIMARY OUTCOMES:
KIT Gene mutation | 15 years
  Number of patients with a molecular analysis positive for KIT mutation
PDGFRA Gene mutation | 15 years
  Number of patients with a molecular analysis positive for PDGFRA mutation
Expression of CD117 | 15 years
  Number of patients with immunohistochemical expression of CD117
Expression of DOG1 | 15 years
  Number of patients with immunohistochemical expression of DOG1
Recurrence | 15 years
  Number of patients with recurrence after treatment with tyrosinkin inhibitors.
Deceased | 15 years
  Number of patients deceased during follow-up.
Location | 15 years
  Location of the tumor (gastric o jejunoileal)

CONTACTS AND LOCATIONS:
Locations (1):
- David Ferreras, Murcia, Spain